CLINICAL TRIAL: NCT00004006
Title: Treatment for Extrachoroidal or Metastatic Retinoblastoma
Brief Title: Combination Chemotherapy, Radiation Therapy, and Bone Marrow Transplantation in Treating Patients With Retinoblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067217; P30CA021765 (NIH); SJCRH: RET4; NCI-G99-1555
Record Dates: First submitted 1999-11-01; First posted 2003-07-18 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma; extraocular retinoblastoma; recurrent retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Topotecan; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: topotecan hydrochloride
Procedure: autologous bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy followed by bone marrow transplantation in treating patients who have retinoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the feasibility of sequential therapy with carboplatin, etoposide, cyclophosphamide, doxorubicin, topotecan and radiotherapy followed by autologous bone marrow transplantation in patients with extrachoroidal or metastatic retinoblastoma.
* Assess this treatment regimen in terms of response and toxicity before and after autologous bone marrow transplantation in this patient population.

OUTLINE: Patients receive carboplatin IV on day 1 and etoposide IV over 1 hour daily on days 1-3 of weeks 0, 6, and 12, plus cyclophosphamide IV or orally daily on days 1-7, doxorubicin IV on day 8 and carboplatin IV over 1 hour on day 10 on weeks 3, 9, and 15. Beginning on week 6, patients receive concurrent radiotherapy 5 days a week over 4-6 weeks. Patients with meningeal involvement receive topotecan intrathecally twice weekly for 3 weeks and then weekly for 3 weeks before starting radiotherapy. Beginning one day after each treatment course, patients receive filgrastim (G-CSF) subcutaneously daily for 10 days.

Patients undergo bone marrow collection before or after week 6. Following hematologic recovery, patients receive several days of high dose chemotherapy consisting of cyclophosphamide and topotecan followed by bone marrow reinfusion.

Patients are followed at 6, 9, and 12 months, and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of extrachoroidal or metastatic retinoblastoma, confirmed by histology, physical examination, or diagnostic imaging

PATIENT CHARACTERISTICS:

Age:

* 15 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy for low stage intraocular disease allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy except to eye(s) or orbit(s)

Surgery:

* Not specified

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 1997-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Rodriguez-Galindo, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org